CLINICAL TRIAL: NCT02285959
Title: Super-Selective Intraarterial Intracranial Infusion of Bevacizumab (Avastin) for Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Global Neurosciences Institute (Other)
Responsible Party: Principal Investigator, Erol Veznedaroglu, MD FAANS FACS FAHA, Global Neurosciences Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GlobalNI
Record Dates: First submitted 2014-11-04; First posted 2014-11-07 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra Arterial Bevacizumab (Experimental): Repeated Intra Arterial bevacizumab injections at 15 mg/kg every 3 weeks
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The high-grade malignant brain tumor glioblastoma multiforme (GBM) comprise the majority of all primary brain tumors in adults. This group of tumors also exhibits the most aggressive behavior, resulting in median overall survival durations of only 9-12 months for GBM. Initial therapy consists of surgical resection, external beam radiation or both. Currently, all patients experience a recurrence after this first-line therapy, so improvements in both first-line and salvage therapy are critical to enhancing quality-of-life and prolonging survival. Superselective Intraarterial Cerebral Infusion (SIACI) is a technique that can effectively increase the concentration of drug delivered to the brain while sparing the body of systemic side effects. This technique threads a tiny catheter through the patient's femoral artery in the leg, up through the body and neck and into the brain. Once the catheter reaches the brain, chemotherapy is released to the blood vessels that feed the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of GBM
* Grade IV GBM tumors that have recurred after total resection
* Age > 18 years
* At least four weeks following any recent surgery
* Patients must have a Karnofsky performance status ≥60% and an expected survival of ≥ three months.
* No IV chemotherapy for three weeks prior to treatment under this research protocol and no external beam radiation for four weeks prior to treatment under this research protocol.
* Patients must have adequate hematologic reserve
* Pre-enrollment coagulation parameters (PT and PTT) must be adequate.
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.
* Patients must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men will be informed as to the potential risk of procreation while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 3 years
  The frequency of adverse events will be quantified until disease progression or death.

SECONDARY OUTCOMES:
Tumor Response | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Philadelphia, Pennsylvania, United States